CLINICAL TRIAL: NCT06556576
Title: e-Intervention Enhancing Mental Health in Adolescents (IMPROVA)
Brief Title: e-Intervention Enhancing Mental Health in Adolescents
Acronym: IMPROVA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Babes-Bolyai University (Other); Linkoeping University (Other Government); Betthera s.r.o. (Other); Wuerzburg University Hospital (Other); University of Ulm (Other); Utrecht University (Other); Ajuntament de Sant Boi de Llobregat (Unknown); VU University of Amsterdam (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Stichting Trimbos-Instituut (Other); University of Deusto (Other); Cliclab Transformative Agent SL (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ORG-100042235
Record Dates: First submitted 2024-07-18; First posted 2024-08-16 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Well-Being, Psychological; Depressive Symptoms; Social Isolation
Keywords: Adolescents; School-based interventions; Health promotion; Mental health
MeSH Terms: conditions — Psychological Well-Being; Depression; Social Isolation

STUDY DESIGN:
Intervention Model Description: The randomization will occur at the country level. Within each country (France, Germany, Romania, and Spain), schools will be randomized to either the intervention or control group. This means that in each country, schools will be assigned to one of the two groups, and all students, their families, teachers, and other school staff within those schools will be placed in the respective group. The same procedure will be followed independently within each of the four countries.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMPROVA intervention group (Experimental): Participants (students, parents, teachers and other school staff) in the IMPROVA group will have access to a series of resources and training with the ultimate goal of promoting mental health and wellbeing among adolescents. This material will be delivered via the IMPROVA platform throughout one school year. IMPROVA platform will be available in app and web-based formats, and participants will be encouraged to utilize it as frequently as possible.
  Interventions: Device: IMPROVA Platform
- CONTROL group (No Intervention): Participants in the control group will not have access to the IMPROVA platform. Their school routine and the support they usually receive will remain unchanged. After the intervention period (school year 2024/25), schools, teachers, school staff, adolescents and their families in the control group will be able to access the IMPROVA platform during the school year 2025/26 (waiting list control group).

INTERVENTIONS:
Device: IMPROVA Platform — Adolescents, teachers, school staff, and parents will have access to a variety of content aimed at promoting the mental health and well-being of adolescents that can be accessed through the IMPROVA platform, an innovative eHealth solution that can be accessed via app and website.
  Students: around 20 modules that can be grouped in five categories: Me and My Emotions, Me and My Body, Me and My Relationships, School and Free time, and Finding my Strengths.
  Teachers and other school staff: 1) pedagogical and health-related modules to support their students and teaching practices; 2) modules to manage their own health; 3) tutoring sessions: resources (lessons plans) for tutors (teachers or other school staff) for carrying out a discussion with students in topics related to the students' health and wellbeing.
  Parents: contents on promoting positive relationships, emotional and social skills, positive behaviour, behaviours to support wellbeing, and family-school collaboration.
  Arms: IMPROVA intervention group

SUMMARY:
The e-Intervention Enhancing Mental Health in Adolescents (IMPROVA) study will co-design, test, evaluate, and facilitate the upscaling of a modular eHealth intervention platform that aims to improve mental health and wellbeing, early detect mental health problems and prevent common mental problems in adolescents. IMPROVA will be implemented in school settings and will include components for adolescents, parents, teachers, and other school staff in complementary and synergistic modules based on materials designed and tested in >20 projects carried out by the consortium members. After alpha, beta and pilot testing of the platform, the IMPROVA program will be implemented via a randomised controlled trial in secondary education schools in France, Germany, Romania and Spain, including approximately 6,000 adolescents. A 360º evaluation of IMPROVA will include Effectiveness, Implementation, Economic, and Social Return on Investment analysis. The primary outcome to assess the effectiveness of the IMPROVA program is the overall mental health of adolescents. A series of secondary outcomes will also evaluate the potential impact of the platform on other health-related outcomes (e.g., wellbeing, social isolation, anxiety, life satisfaction). Using implementation science methodology, IMPROVA will co-design transferable evidence-based guidance for scaling up the platform with users and policymakers. IMPROVA aims to provide an evidence-based, innovative, large-scale, comprehensive intervention, and a scale-up plan to promote mental health and prevent mental disorders in adolescents; empower adolescents and families to make better decisions regarding their mental health; and provide schools and the community with tools to achieve a society with better mental health and lower stigma.

DETAILED DESCRIPTION:
The e-Intervention Enhancing Mental Health in Adolescents (IMPROVA) study's main objective is to co-design, test and facilitate the upscaling of a modular eHealth intervention platform that aims to improve mental health and wellbeing, early detect mental health problems and prevent common mental problems in adolescents.

The IMPROVA program is a universal intervention to be implemented in school settings and will include components for adolescents, parents, teachers, and other school staff. Therefore, teachers and other school staff working in secondary schools in France, Germany, Romania and Spain together with enrolled students and their parents will be invited to access the intervention content via an eHealth platform - The IMPROVA platform.

Users will be able to access the contents via an app or web browser. Each user type will have access to content specifically tailored for them, with the ultimate goal of promoting mental health and wellbeing among adolescents.

* Students will have access to around 20 modules that can be grouped into five categories: Me and My Emotions, Me and My Body, Me and My Relationships, Schools and Free time, and Finding my Strengths.
* Teachers and other school staff will have access to pedagogical and health-related modules aiming to support their students and teaching practices (Supporting students), and to modules to manage their health (My own health). In addition, the tutoring sessions are resources (lessons plans) for tutors (teachers or other school staff) for carrying out a discussion with students in topics related to the students' health and wellbeing.
* Parents will have access to content on promoting positive relationships, emotional and social skills, positive behaviour, behaviours to support wellbeing, and family-school collaboration.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents enrolled in the selected secondary schools will be eligible.
* Parents of adolescents enrolled in the selected schools will be eligible
* Teachers and school staff: All teachers and school staff working in the selected schools will be eligible.
* Participants can be of any gender.
* Teachers and school staff will have to be older than 18 years.

Exclusion Criteria:

• Apart from not signing the informed consent, no exclusion criteria will be applied.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Strengths and Difficulties Questionnaire (SDQ) | Baseline (pre-intervention), mid-term evaluation (during the intervention), post-intervention (immediately after the intervention), and follow up (13-14 months after baseline)
  The SDQ is a brief behavioural screening questionnaire for children and adolescents, typically used to assess various aspects of their behaviour and emotions. It consists of 25 items, divided into five subscales:
  * Emotional Symptoms
  * Conduct Problems
  * Hyperactivity/Inattention
  * Peer Relationship Problems
  * Prosocial Behavior
  Change in the score of the Strengths and Difficulties Questionnaire that ranges from 0 to 40 points (sum of four subscales: Emotional Symptoms, Conduct Problems, Hyperactivity/Inattention, and Peer Relationship Problems). A higher score indicates a poorer overall mental health.
  The total score can also be interpreted in the following categories:
  Normal: 0-13 Borderline: 14-16 Abnormal: 17-40
  The Prosocial Behaviour Subscale score ranges from 0 to 10, and is interpreted separately:
  Normal: 6-10 Borderline: 5 Abnormal: 0-4

SECONDARY OUTCOMES:
KIDSCREEN-10 | Baseline (pre-intervention), mid-term evaluation (during the intervention), post-intervention (immediately after the intervention), and follow up (13-14 months after baseline)
  KIDSCREEN-10 has 10 items and measures general health-related quality of life (HRQoL) for adolescents.
  Scoring: Each item on the KIDSCREEN-10 is rated on a 5-point Likert scale, reflecting the frequency or intensity of the feelings or behaviours described. The scores for the 10 items are summed to produce a total score. This total score can then be transformed into a T-score or percentile rank, based on normative data, to facilitate interpretation. The higher the total score, the better the reported HRQoL.
Goal-Based Outcome Measure (GBO) | Baseline (pre-intervention), mid-term evaluation (during the intervention), post-intervention (immediately after the intervention), and follow up (13-14 months after baseline)
  It is a method used to assess treatment progress and outcomes based on specific goals set by the adolescent. It is designed to capture changes in individuals' functioning and well-being that are meaningful and relevant to them, rather than relying solely on standardized symptom measures.
  Adolescents will be asked to select three goals they would like to achieve by the end of the current school year, and on a scale from 0 to 10, choose the number that best describes how close they are to reaching their goal on that moment (0 means no progress has been made towards a goal, a score of 10 means a goal has been reached fully).
PHQ-8 | Baseline (pre-intervention), mid-term evaluation (during the intervention), post-intervention (immediately after the intervention), and follow up (13-14 months after baseline)
  The PHQ-8 consists of 8 items that correspond to the diagnostic criteria for major depressive disorder (MDD) in the DSM-IV and DSM-5. Each item addresses a specific symptom of depression and is rated based on the frequency of the symptom over the past two weeks.
  Scoring: Each of the 8 items is rated on a 4-point scale. The total score ranges from 0 to 24. The total score is used to determine the severity of depression: 0-4: Minimal or none, 5-9: Mild, 10-14: Moderate, 15-19: Moderately severe, 20-24: Severe
GAD-7 | Baseline (pre-intervention), mid-term evaluation (during the intervention), post-intervention (immediately after the intervention), and follow up (13-14 months after baseline)
  The GAD-7 consists of 7 items that correspond to the diagnostic criteria for GAD. Each item asks about the frequency of anxiety-related symptoms over the past two weeks.
  Scoring: Each of the 7 items is rated on a 4-point scale. The total score ranges from 0 to 21. The total score is used to determine the severity of anxiety: 0-4: Minimal anxiety, 5-9: Mild anxiety, 10-14: Moderate anxiety, 15-21: Severe anxiety
Social isolation questionnaire | Baseline (pre-intervention), mid-term evaluation (during the intervention), post-intervention (immediately after the intervention), and follow up (13-14 months after baseline)
  The Social isolation questionnaire is composed of 17 items that can be categorised into three domain: feelings of loneliness, friendships, and family support.
  Scoring: score can assume values from 0 to 131, with 0 characterizing an adolescent with a minimum score of social isolation, and 131 an adolescent with a maximum score of social isolation.
Teachers and Classmate Support Scale | Baseline (pre-intervention), post-intervention (immediately after the intervention), and follow up (13-14 months after baseline)
  It is a measure designed to assess the perceived support that students receive from their teachers and classmates.
  It consists of two subscales: Teacher Support and classmate support.
  Scoring: For each subscale, the scores for the individual items (1 to 5) are summed to obtain a total score (3-15). Higher scores indicate higher perceived support from teachers or classmates.
Cantril Ladder Scale | Baseline (pre-intervention), mid-term evaluation (during the intervention), post-intervention (immediately after the intervention), and follow up (13-14 months after baseline)
  The Cantril Ladder Scale consists of a visual representation of a ladder with steps numbered from 0 at the bottom to 10 at the top. Adolescents will be asked to imagine that the ladder represents their life in two scenarios: 1) The Present Life Evaluation, and 2) Future Life Expectations
  The top of the ladder (step 10) represents the "best possible life" they could imagine.
  The bottom of the ladder (step 0) represents the "worst possible life" they could imagine.
Single-Item Self-Esteem Scale (SISE) | Baseline (pre-intervention), mid-term evaluation (during the intervention), post-intervention (immediately after the intervention), and follow up (13-14 months after baseline)
  It is a brief self-report measure designed to assess adolescent's overall self-esteem with a single question.
  Adolescents will rate their overall self-esteem on a scale ranging from 1 to 7, with higher numbers indicating higher self-esteem.
Revised Self-theory Scale | Baseline (pre-intervention), post-intervention (immediately after the intervention), and follow up (13-14 months after baseline)
  The Revised Self-theory Scale is a 8-item scale to assess adolescents' beliefs about themselves in relation to their ability to change their mindsets (Fixed or Growth mindset).
  Scoring: Likert scale ranging from 1-strongly disagree to 6 strongly agree. The total score range from 8 to 48. The higher the score, the more a fixed mindset, the lower the score, the more of a growth mindset.
15-item School Engagement Scale | Baseline (pre-intervention), post-intervention (immediately after the intervention), and follow up (13-14 months after baseline)
  The 15-item School Engagement Scale (SES) is a self-report measure used to assess various dimensions of student engagement in the school environment. Developed to capture students' psychological investment in learning and academic activities, the SES evaluates multiple facets of engagement that contribute to positive educational outcomes.
  Scoring: Scores on the SES are calculated by summing the responses across all items or within specific subscales (Behavioural, Emotional, Cognitive ). Higher scores indicate greater levels of engagement in the respective dimension.
Revised Bully/Victim Questionnaire | Baseline (pre-intervention), post-intervention (immediately after the intervention), and follow up (13-14 months after baseline)
  Revised Bully/Victim Questionnaire is a four-item questionnaire to assess to which extend the adolescent engaged or was a victim of bullying/cyberbullying. The items can be answered (and scored) in a 5-point Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Josep Maria Haro, PhD, Principal Investigator — Fundació Sant Joan de Déu

IPD SHARING:
Plan to Share IPD: Yes
The e-Intervention Enhancing Mental Health in Adolescents (IMPROVA) study plans to make IPD available, but the concrete plan is not defined yet. IMPROVA will follow the FAIR criteria for research data, and make, at least partially, the research data Findable, Accessible, Interoperable and Re-usable (FAIR).
  The plan is that third parties (e.g., other researchers) might get access to the IMPROVA anonymised/pseudoanonymised data, however, after a certain embargo period. This embargo period will give the consortium the opportunity to exploit the dataset herself, before allowing others to use the collected data.
Time Frame: The Intellectual Property and Dissemination Board (IPDB) of the project will still establish the exact duration of the embargo and this might vary for the different datasets.
Access Criteria: The procedure for data access by third parties will be in accordance with the procedure to be stablished by the Intellectual Property and Dissemination Board of the project.